CLINICAL TRIAL: NCT00597519
Title: A Myeloablative Conditioning Regimen Consisting of Cyclophosphamide, Fludarabine and Total Body Irradiation Followed by the Transplantation of Unrelated Donor Double Unit Umbilical Cord Blood Grafts for Patients With Hematological Malignancy.
Brief Title: A Myeloablative Conditioning Regimen and Total Body Irradiation Followed by the Transplantation for Patients With Hematological Malignancy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-014; CA23766; NCT00388102 (obsolete NCT alias)
Record Dates: First submitted 2007-12-26; First posted 2008-01-18 (Estimated); Results first posted 2016-02-12 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-01

CONDITIONS: Cancer; Leukemia; Myelodysplastic Syndrome; Non-Hodgkin's Lymphoma
Keywords: Cancer; Leukemia; Myelodysplastic Syndrome; Non-Hodgkin's Lymphoma; Total Body Irradiation; Umbilical Cord Blood Grafts; 06-014
MeSH Terms: conditions — Neoplasms; Leukemia; Myelodysplastic Syndromes; Lymphoma, Non-Hodgkin | interventions — fludarabine; Cyclophosphamide; Transplantation

ARMS (1):
- Treatment (Experimental): Patients with hematopoietic malignancy at high-risk for relapse or with advanced disease will receive myeloablative conditioning with cyclophosphamide (Cy), low dose fludarabine (Flu) and total body irradiation (TBI) with post transplantation cyclosporine (CSA) and mycophenolate mofetil (MMF) for GVHD prophylaxis.
  Interventions: Drug: Fludarabine, Cyclophosphamide; Procedure: Transplantation

INTERVENTIONS:
Drug: Fludarabine, Cyclophosphamide — Fludarabine 25 mg/m2/day IV in the morning x 3 days (days -7, -6 and -5) for a total dose of 75 mg/m2 followed by Cyclophosphamide on days -6 and -5. 60mg/kg/day IV over 30-60 minutes x 2 days (days -6 and -5). High volume fluids should commence approximately 12 hours prior to drug and continue until 24 hours after second dose.
  Total Body Irradiation: 125 cGy x 11 doses (TID on days -3, -2, -1 and BID on day 0) for a total TBI dose of 1375 cGy. Pediatric patients unable to tolerate a TID dosing schedule can receive 150 cGy x 8 doses (BID on days -3, -2, -1, and 0). All patients will receive GVHD prophylaxis with 2 drugs: Cyclosporine A and Mycophenolate mofetil (MMF).
  Units should be given consecutively each over approximately 10-30 minutes.Pre-medication should include acetaminophen and diphenhydramine or hydroxyzine.G-CSF 5 mcg/kg/day IV/SQ (dose rounded to vial size to a maximum of 480 mcg) will be given from day +1 until ANC recovery.
Procedure: Transplantation — The UCB ( Umbilical Cord Blood) collection known as a unit is processed to remove excess plasma and red cells, tested for sterility, HLA-typed, cryopreserved and stored. This protocol involves the administration of two UCB units from two different donors. The units will be thawed in the Cytotherapy Laboratory as per the current standard operating procedure.

SUMMARY:
In this study two cord blood collections will be used to increase the number of cord blood cells you will receive on transplant day. We call this a "double unit" cord blood transplant. A previous study suggests double unit cord blood transplant may have a better result. The main purpose of this study is to find out how good a cord blood transplant using two cord blood collections from two different babies is at curing you of your cancer. Double unit cord blood transplants are now being studied as a way to increase the number of cord blood cells given to bigger children and adult patients.

Based on studies that have already been done double unit cord blood transplant appears to be safer than if only one cord blood unit is used. However, double unit cord blood transplant is a fairly new form of treatment.

DETAILED DESCRIPTION:
This is a single arm phase 2 study to obtain a preliminary estimate of efficacy of myeloablative double unit umbilical cord blood transplantation (UCBT) as measured by overall and disease-free survival at 1 year post transplantation. The UCB graft will consist of two (or double) units from two unrelated newborn donors. Patients with hematopoietic malignancy at high-risk for relapse or with advanced disease will receive myeloablative conditioning with cyclophosphamide (Cy),low dose fludarabine (Flu) and total body irradiation (TBI) with post transplantation cyclosporine (CSA) and mycophenolate mofetil (MMF) for GVHD prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* Age 4 - 50 years
* Patient should not have a related or unrelated volunteer donor that is suitably HLA matched and available in the required time period or be a suitable candidate for an autologous stem cell transplant.
* Patients will have one of the following hematological malignancies: Acute myelogenous leukemia (AML):

  * Complete first remission (CR1) at high risk for relapse as defined by:

known prior diagnosis of myelodysplasia (MDS); or therapy related AML; or White cell count at presentation > 100,000; or Presence of extramedullary leukemia at diagnosis; or Unfavorable FAB type (M0, M5-7); or High-risk cytogenetics (such as those associated with MDS, abnormalities of 5, 7, 8, Philadelphia chromosome, complex karyotype); or High risk molecular markers such as FLT3 mutations; or Requirement for 2 or more inductions to achieve CR1

* Complete second CR (CR2).

  • Acute lymphoblastic leukemia (ALL):
* Complete first remission (CR1) at high risk for relapse as defined by:

White cell count at presentation as follows:

* > 100,000 if < 18 years
* > 50,000 if > 18 years; or

Presence of extensive extra-medullary disease (excluding CNS disease); or Presence of high-risk cytogenetic abnormality such as t(9;22), t(1;19), t(4;11) or other MLL rearrangements (11q23), t(8;14) [excluding B-ALL in pediatric patients]; or

Failed to achieve complete remission after four weeks of induction therapy Unable to receive required consolidation chemotherapy as would be needed to maintain remission

* Complete second or third remission (CR2 or CR3)

  * Acute undifferentiated leukemia (AUL), infant leukemia, or biphenotypic leukemia in CR1, CR2 or CR3. Patients with infant leukemia must be eligible to receive total body irradiation.
  * Juvenile Myelomonocytic leukemia (JMML) with < 30% bone marrow blasts.
  * Chronic myelogenous leukemia (CML)
* GleevecTM failure in 1st or 2nd chronic phase;
* Gleevec failure in 1st or 2nd accelerated phase.

  • Myelodysplastic Syndrome (MDS) with one of the following:
* Low (Score 0) International Prognostic Scoring System (IPSS) score with Life-threatening cytopenia(s); or Red cell or platelet transfusion dependent
* Intermediate (Score 1) or High (Score 2) International Prognostic Scoring System (IPSS) score.
* Patients with bone marrow blasts > 10% should have AML induction therapy with disease response to < 5% blasts and at least partial count recovery.

  • Non-Hodgkin's Lymphoma
* Patients with high-grade disease following initial therapy and are not appropriate for further chemotherapy or autologous stem cell transplantation.
* Patients with high-grade or diffuse large cell NHL with recurrent disease after first remission and must have:

Chemo-sensitivity as evidenced by > partial remission (PR) (defined as > 50% reduction in mass size after therapy).

* Patients with adequate organ function and performance status criteria as measured by:
* Karnofsky score > or = to 70 % or Lansky score > or = to 70%
* Renal: Calculated creatinine clearance > or = to 60 ml/min
* Hepatic: Total bilirubin < 2.5 mg/dL unless benign congenital hyperbilirubinemia (Gilbert's syndrome) and ALT/AST < 3 x upper limit of normal
* Albumin > or = to 2.5
* Pulmonary: Pulmonary function (spirometry and corrected DLCO) > or = to 60% normal if available (in small children use History and Physical and CT scan as necessary to determine pulmonary status)
* Cardiac: Left ventricular ejection fraction > or = to 50%
* Double Unit Umbilical Cord Blood Grafts:

Units will be selected based on the HLA match to the patient and on the basis of the individual and combined cell doses of the units.

* Patient has a related or unrelated volunteer donor that is suitably HLA matched and available in the required time period.
* Patient is a candidate for an autologous stem cell transplant.
* Active CNS leukemia.
* Acute Myelogenous Leukemia in greater than CR2.
* Acute Myelogenous Leukemia evolved from myelofibrosis.
* Acute Lymphoblastic Leukemia, acute undifferentiated leukemia, biphenotypic leukemia or infant leukemia greater than CR3.
* Any acute leukemia with:

  * Morphologic relapse or persistent disease in the BM (cytogenetic relapse without morphologic evidence of relapse or cytogenetic persistent disease in the BM is acceptable); or
  * Active extra-medullary leukemia; or
  * Requiring greater than 2 cycles of chemotherapy to obtain present remission status;
* Bone Marrow aplasia (defined as BM cellularity less than 5% at transplant work-up); or
* MDS with greater than 10% bone marrow blasts refractory to chemotherapy; or
* CML in blast crisis; or
* NHL refractory to chemotherapy (less than PR after 2 or more regimens); or
* Prior autologous or allogeneic HSC transplant at any time; or
* Prior radiation therapy rendering patient ineligible for TBI; or
* Uncontrolled viral, bacteria or fungal infection at time of study enrollment; or
* Seropositive or NAT positive for HIV; or
* Females who are pregnant or breast feeding; or
* Patient or guardian unable to give informed consent or unable to comply with the treatment protocol including appropriate supportive care, follow-up, and research tests.

Ages: 4 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2006-03; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juliet Barker, MBBS, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering web site — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: Cyclophosphamide, Fludarabine and Total Body Irradiation Followed by the Transplantation of Unrelated Donor Double Unit Umbilical Cord Blood Grafts for Patients with Hematological Malignancy
Period: Overall Study
Arm/Group | Treatment
Started | 28
Completed | 27
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16
  Between 18 and 65 years | 12
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Overall Response
Description: To obtain a preliminary estimate of efficacy of double unit UCBT as measured by overall response.
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 27
participants
  Complete Remission | 24
  Relapse | 3

ADVERSE EVENTS:
Arm/Group | Treatment
Serious Adverse Events (participants affected / at risk) | 8/28
Other Adverse Events (participants affected / at risk) | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=28)
Blood/Bone Marrow, other (Blood and lymphatic system disorders) | 1
Death not associated with CTCAE term- Death NOS (General disorders) | 4
Death not associated with CTCAE term- Sudden death (General disorders) | 1
Death not associated with CTCAE term-Disease progression NOS (General disorders) | 2
Pain - Abdomen NOS (General disorders) | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=28)
Albumin, low (hypoalbuminemia) (Metabolism and nutrition disorders) | 2
Alkaline phosphatase (Metabolism and nutrition disorders) | 2
ALT, SGPT (Blood and lymphatic system disorders) | 11
Amylase (Blood and lymphatic system disorders) | 3
AST, SGOT (Blood and lymphatic system disorders) | 9
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 10
Creatinine (Metabolism and nutrition disorders) | 2
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 16
Hemoglobin (Blood and lymphatic system disorders) | 28
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 28
Lipase (Metabolism and nutrition disorders) | 2
Lymphopenia (Blood and lymphatic system disorders) | 28
Magnesium, high (hypermagnesemia) (Metabolism and nutrition disorders) | 11
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 28
Phosphate, low (hypophosphatemia) (Metabolism and nutrition disorders) | 7
Platelets (Blood and lymphatic system disorders) | 28
Potassium, high (hyperkalemia) (Metabolism and nutrition disorders) | 8
Potassium, low (hypokalemia) (Metabolism and nutrition disorders) | 15
PTT (Blood and lymphatic system disorders) | 5
Sodium, low (hyponatremia) (Metabolism and nutrition disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes